CLINICAL TRIAL: NCT01512108
Title: A 52-week, Multi-centre, Open-labelled, Randomised (2:1), Parallel-group Trial With an Active Control (Two OADs Combination Therapy) to Evaluate the Safety and Efficacy of Liraglutide in Combination With an OAD in Subjects With Type 2 Diabetes Insufficiently Controlled on OAD Monotherapy
Brief Title: Safety and Efficacy of Liraglutide in Combination With an OAD in Subjects With Type 2 Diabetes Insufficiently Controlled on OAD Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-3924; U1111-1121-3457 (Other: WHO); JapicCTI-121744 (Registry Identifier: JAPIC)
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide + an OAD therapy (Experimental)
  Interventions: Drug: liraglutide
- Two OADs combination therapy (Active Comparator)
  Interventions: Drug: oral anti-diabetic drug

INTERVENTIONS:
Drug: liraglutide — 0.9 mg/day liraglutide was injected once daily subcutaneously (s.c., under the skin).
  Arms: Liraglutide + an OAD therapy
Drug: oral anti-diabetic drug — An additional oral anti-diabetic drug (OAD) with a different mechanism of action than the pre-trial OAD. The type and dosage of the additional OAD should be chosen by the investigator within the Japanese labelled dose.
  Arms: Two OADs combination therapy

SUMMARY:
This trial was conducted in Japan. The aim of this trial was to evaluate the safety and efficacy of once daily administration of liraglutide in combination with an oral anti-diabetic drug (OAD) in Japanese subjects with type 2 diabetes who are insufficiently controlled on OAD monotherapy. All subjects will continue their pre-trial OAD (either glinide, metformin, alpha-glucosidase inhibitor or thiazolidinedione) during the trial at unchanged type and dose.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject.)
* Japanese subjects with type 2 diabetes on monotherapy with an OAD (either glinide, metformin, a-glucosidase inhibitor or thiazolidinedione) within approved Japanese labelling in addition to diet and exercise therapy. Total daily dose and type of drug should have remained unchanged for at least 8 weeks prior to Visit 1
* Type 2 diabetes mellitus (clinically diagnosed) for at least 6 months
* HbA1c between 7.0-10.0% (both inclusive)
* Body Mass Index (BMI) below 40.0 kg/m^2
* Outpatients who have no plans for an educational hospitalisation for the purpose of glycaemic control. However, hospitalisation for training of self-injection from Visit 2 that is for no longer than one week is allowed
* Subjects able and willing to perform self-monitoring of plasma glucose (SMPG)

Exclusion Criteria:

* Subjects with known or previous malignant tumor and are strongly suspected of recurrence (except basal cell skin cancer or squamous cell skin cancer)
* Calcitonin above or equal to 160 pg/mL
* Personal history of non-familial medullary thyroid carcinoma
* Family or personal history of multiple endocrine neoplasia type 2 (MEN-2) or familial medullary thyroid carcinoma (FMTC)
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Treatment with GLP-1 receptor agonist or dipeptidyl peptidase 4 (DPP-4) inhibitor within 12 weeks prior to Visit 1
* Having contraindications to liraglutide and any of the OADs (according to Japanese labelling)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2013-04-26 (Actual); Study Completion 2013-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (29):
- Japan (29):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ehime, Japan
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Fukuoka, Japan
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Kamagaya-shi, Chiba
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Kurume-shi, Fukuoka
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tagajō-shi
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yamaguchi
  - Novo Nordisk Investigational Site, Yokohama

REFERENCES:
- [Result] Kaku K, Kiyosue A, Ono Y, Shiraiwa T, Kaneko S, Nishijima K, Bosch-Traberg H, Seino Y. Liraglutide is effective and well tolerated in combination with an oral antidiabetic drug in Japanese patients with type 2 diabetes: A randomized, 52-week, open-label, parallel-group trial. J Diabetes Investig. 2016 Jan;7(1):76-84. doi: 10.1111/jdi.12367. Epub 2015 Jul 14. PMID 26816604
- [Result] Kiyosue A, Seino Y, Nishijima K, Bosch-Traberg H, Kaku K. Safety and efficacy of the combination of the glucagon-like peptide-1 receptor agonist liraglutide with an oral antidiabetic drug in Japanese patients with type 2 diabetes: Post-hoc analysis of a randomized, 52-week, open-label, parallel-group trial. J Diabetes Investig. 2018 Jul;9(4):831-839. doi: 10.1111/jdi.12759. Epub 2017 Nov 24. PMID 28984041
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 36 sites in Japan.
Groups:
- Liraglutide 0.9 mg/Day: Liraglutide 0.9 mg/day was injected subcutaneously, once daily in morning or evening in addition to unchanged pre-trial oral anti-diabetic drug (OAD) (either glinide, metformin, α-glucosidase inhibitor or thiazolidinedione) for 52 weeks. Liraglutide was started at 0.3 mg/day and dose was escalated to maximum dose level of 0.9 mg/day by weekly increment of 0.3 mg.
- Additional OAD: Subject's received additional OAD to pre-trial OAD. The type and dosage of additional OAD was chosen based on each individual's glycaemic control by the investigator as per Japanese labelling.
Period: Overall Study
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Started | 243 | 120
Exposed | 240 (3 subjects withdrew prior to exposure to trial drug) | 120
Completed | 221 | 111
Not Completed | 22 | 9
Not completed — Adverse Event | 9 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal Criteria | 1 | 0
Not completed — Unclassified | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD | Total
Number analyzed (Participants) | 240 | 120 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (11.6) | 59.2 (10.2) | 59.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 40 | 98
  Male | 182 | 80 | 262
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.1 (0.8) | 8.1 (0.8) | 8.1 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.68 (1.61) | 8.96 (1.82) | 8.77 (1.69)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (AEs)
Description: Adverse events were defined as events occurring after administration of trial product and no later than 7 days after last day of treatment. Severe AEs: considerable interference with subject's daily activities. Moderate AEs: Marked symptoms, moderate interference with the subject's daily activities. Mild AEs: No or transient symptoms, no interference with the subject's daily activities. Serious AEs: AEs that resulted in any of the following: death, a life-threatening experience, hospitalization/prolongation of existing hospitalization, persistent/significant disability, and congenital anomaly.
Time Frame: Week 0 to Week 52 + 7 days
Population: Safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Number analyzed (Participants) | 240 | 120
Events/100 years of patient exposure
  All AEs | 361 | 331
  Mild AEs | 345 | 321
  Moderate AEs | 14 | 9
  Severe AEs | 2 | 2
  Serious AEs | 5 | 9

2. Secondary Outcome: Number of Confirmed Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes consisted of the pool of episodes of severe hypoglycaemia as well as minor hypoglycaemic episodes [An episode with symptoms consistent with hypoglycaemia with confirmation by plasma glucose <3.1 mmol/L (56 mg/dL) or full blood glucose <2.8 mmol/L (50 mg/dL) and which is handled by the subject himself or herself or any asymptomatic PG value <3.1 mmol/L (56 mg/dL) or full blood glucose value <2.8 mmol/L (50 mg/dL)] with a confirmed plasma glucose value of less than 3.1 mmol/L (56 mg/dL).
Time Frame: Week 0 to Week 52
Population: Safety analysis set includes all subjects who received at least one dose of the trial product.
Measure: Number; unit: episodes
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Number analyzed (Participants) | 240 | 120
episodes | 7 | 2

3. Secondary Outcome: Change in HbA1c From Baseline to Week 52
Description: Estimated mean change in HbA1c from baseline after 52 Weeks of treatment
Time Frame: Week 0, week 52
Population: Full analysis set (FAS) included all randomised subjects who received at least one dose of trial products and missing data were imputed using last observation carried forward (LOCF). One subject did not contribute to the statistical analysis at Week 52.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Number analyzed (Participants) | 239 | 120
percentage of glycosylated haemoglobin | -1.21 (0.05) | -0.94 (0.07)
Statistical Analysis 1: Comparison: Liraglutide 0.9 mg/Day vs Additional OAD; Test type: Superiority or Other; p = 0.0026, ANOVA; Estimated treatment difference, Mean = -0.27, 95% CI [-0.44 to -0.09]

4. Secondary Outcome: Change in FPG From Baseline to Week 52
Description: Estimated mean change from baseline in FPG after 52 Weeks of treatment
Time Frame: Week 0, week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Number analyzed (Participants) | 239 | 120
mmol/L | -1.55 (0.09) | -1.24 (0.12)
Statistical Analysis 1: Comparison: Liraglutide 0.9 mg/Day vs Additional OAD; Test type: Superiority or Other; p = 0.0458, ANOVA; Estimated treatment difference, Mean = -0.30, 95% CI [-0.60 to -0.01]

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of consent until 52 weeks of treatment and if needed were followed up after the final visit.
Description: Safety analysis set included all subjects who received at least one dose of the trial product.
Arm/Group | Liraglutide 0.9 mg/Day | Additional OAD
Serious Adverse Events (participants affected / at risk) | 11/240 | 10/120
Other Adverse Events (participants affected / at risk) | 161/240 | 77/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.9 mg/Day (N=240) | Additional OAD (N=120)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Meningitis herpes (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide 0.9 mg/Day (N=240) | Additional OAD (N=120)
Cataract (Eye disorders) | 8 (8) | 8 (8)
Diabetic retinopathy (Eye disorders) | 21 (22) | 16 (16)
Abdominal discomfort (Gastrointestinal disorders) | 19 (21) | 1 (1)
Constipation (Gastrointestinal disorders) | 44 (48) | 12 (13)
Dental caries (Gastrointestinal disorders) | 7 (7) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 20 (25) | 9 (10)
Nausea (Gastrointestinal disorders) | 31 (33) | 4 (4)
Influenza (Infections and infestations) | 8 (8) | 6 (6)
Nasopharyngitis (Infections and infestations) | 89 (135) | 47 (85)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 3 (3)
Headache (Nervous system disorders) | 12 (14) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.